CLINICAL TRIAL: NCT03957837
Title: Optical Nerve Sheath Diameter Changes During Steep Trendelenburg Position for Laparoscopic Prostatectomy
Brief Title: Optical Nerve Sheath Changes During Head Down Laparoscopy
Status: Completed | Type: Observational
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Riccardo Colombo, Principal Investigator, ASST Fatebenefratelli Sacco
Other Study IDs: RIA02/2019
Record Dates: First submitted 2019-05-19; First posted 2019-05-21 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Intracranial Hypertension; Brain Edema; Pneumoperitoneum; Surgery, Laparoscopic
MeSH Terms: conditions — Intracranial Hypertension; Brain Edema; Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Steep Trendelenburg: Patients undergoing elective laparoscopic prostatectomy in steep Trendelenburg position (25 degrees head down position)
  Interventions: Diagnostic Test: Optical nerve sheath diameter ultrasound measurement
- Healthy controls: Healthy awake volunteers undergoing steep Trendelenburg position (25 degrees head down position)
  Interventions: Diagnostic Test: Optical nerve sheath diameter ultrasound measurement

INTERVENTIONS:
Diagnostic Test: Optical nerve sheath diameter ultrasound measurement — In cases: ultrasound measurement of the diameter of the optical nerve sheath at (T1) baseline before the induction of general anesthesia (5 min after the beginning of mechanical ventilation in supine position); (T2) after 10 min from 25 degrees head down positioning and with pneumoperitoneum insufflation; (T3) after 60 min from T2, in head down position; (T4) after 10 min from tracheal tube removal, in supine position.
  In healthy controls: ultrasound measurement of the diameter of the optical nerve sheath at (T1) baseline in supine position; (T2) after 10 min from 25 degrees head down positioning; (T3) after 60 min from T2, in a head down position; (T4) after 10 min from positioning supine

SUMMARY:
Patient undergoing laparoscopic radical prostatectomy in steep trendelenburg position are at risk to develop complication from brain edema.

Ultrasound assessment of optical nerve sheath diameter is a simply, non-invasive method to estimate the increase of intracranial pressure. It is unknown how optical nerve sheath diameter changes after prolonged head down position.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective laparoscopic prostatectomy in steep Trendelenburg position
* American Society of Anesthesiologists risk I-III

Exclusion Criteria:

* Age <18 or >70 years
* American Society of Anesthesiologists risk >III
* Assumption of beta-2-blockers, diuretics
* Heart failure with NYHA class ≥ IIb
* Diabetes with ocular (i.e. retinopathy), neurologic (i.e. peripheral neuropathy), or renal complications
* History of cardiac surgery, thoracic surgery, suprainguinal vascular surgery, head surgery, ocular surgery, stroke, hydrocephalus.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective laparoscopic radical prostatectomy
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Optical nerve sheath diameter changes during steep Trendelenburg position | 2 months
  changes of optical nerve sheath diameter in millimeters measured by ultrasound in patients undergoing laparoscopic radical prostatectomy and in healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Fatebenefratelli Sacco, Luigi Sacco Hospital, Milan, Italy

REFERENCES:
- [Background] Guillonneau B, Cathelineau X, Barret E, Rozet F, Vallancien G. Laparoscopic radical prostatectomy: technical and early oncological assessment of 40 operations. Eur Urol. 1999;36(1):14-20. doi: 10.1159/000019921. PMID 10364650
- [Background] Gainsburg DM, Wax D, Reich DL, Carlucci JR, Samadi DB. Intraoperative management of robotic-assisted versus open radical prostatectomy. JSLS. 2010 Jan-Mar;14(1):1-5. doi: 10.4293/108680810X12674612014266. PMID 20529522
- [Background] Halverson A, Buchanan R, Jacobs L, Shayani V, Hunt T, Riedel C, Sackier J. Evaluation of mechanism of increased intracranial pressure with insufflation. Surg Endosc. 1998 Mar;12(3):266-9. doi: 10.1007/s004649900648. PMID 9502709
- [Background] Awad AA, Ghobashy MA, Ouda W, Stout RG, Silverman DG, Shelley KH. Different responses of ear and finger pulse oximeter wave form to cold pressor test. Anesth Analg. 2001 Jun;92(6):1483-6. doi: 10.1097/00000539-200106000-00026. PMID 11375830
- [Background] Dubourg J, Javouhey E, Geeraerts T, Messerer M, Kassai B. Ultrasonography of optic nerve sheath diameter for detection of raised intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2011 Jul;37(7):1059-68. doi: 10.1007/s00134-011-2224-2. Epub 2011 Apr 20. PMID 21505900